CLINICAL TRIAL: NCT07273136
Title: Safety and Efficacy of Combined Subcostal and Lateral Transversus Abdominis Plane Block for Postoperative Analgesia Versus Thoracic Epidural Analgesia in Patients Undergoing Major Abdominal Cancer Surgery
Brief Title: Combined Subcostal and Lateral Transversus Abdominis Plane Block for Postoperative Analgesia Versus Thoracic Epidural Analgesia in Patients Undergoing Major Abdominal Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaa Gamal Saad Mohamed, Anesthesia and Intensive Care, Faculty of Medicine, Assiut University, Assiut, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 620
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Subcostal; Lateral; Transversus Abdominis Plane Block; Postoperative Analgesia; Thoracic Epidural Analgesia; Major Abdominal Cancer Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcostal and lateral transversus abdominis plane block group (Experimental): Patients will receive an ultrasound-guided combined subcostal and lateral transversus abdominis plane block.
  Interventions: Other: Subcostal and lateral transversus abdominis plane block
- Thoracic epidural anesthesia group (Active Comparator): Patients will receive an ultrasound-guided thoracic epidural anesthesia.
  Interventions: Other: Thoracic epidural anesthesia

INTERVENTIONS:
Other: Subcostal and lateral transversus abdominis plane block — Patients will receive an ultrasound-guided combined subcostal and lateral transversus abdominis plane block.
  Arms: Subcostal and lateral transversus abdominis plane block group
Other: Thoracic epidural anesthesia — Patients will receive an ultrasound-guided thoracic epidural anesthesia.
  Arms: Thoracic epidural anesthesia group

SUMMARY:
This study aims to evaluate the safety and efficacy of combined subcostal and lateral transversus abdominis plane (TAP) for postoperative analgesia versus thoracic epidural anesthesia (TEA) in patients undergoing major abdominal cancer surgery.

DETAILED DESCRIPTION:
Postoperative pain is treated using a variety of techniques. It is possible to deliver opioids intravenously, neuraxially, or both.

Thoracic epidural anesthesia (TEA) has long been considered the benchmark for analgesia in major abdominal operations due to its consistent efficacy in pain control and additional benefits such as reduced ileus and improved pulmonary function.

Transversus abdominis plane (TAP) blocks can be a critical component of postoperative pain management, and they play a crucial role in Enhanced Recovery After Surgery (ERAS) protocols, as they significantly affect recovery and patient well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Scheduled for major abdominal surgeries including: (e.g., gastrectomy, colectomy, hepatectomy, cystectomy, total abdominal hysterectomy, Nephrectomy, pancreatectomy).

Exclusion Criteria:

* Intraoperative hemodynamic instability.
* History or evidence of coagulopathy.
* Infection or abdominal wall masses at injection site.
* Morbid obesity.
* Other Medical conditions including mental illness or substance abuse.
* Known allergy to local anesthetics.
* Chronic opioid use or chronic pain conditions.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the Visual Analogue Scale (VAS) > 3 to be repeated after 30 min if pain persists until the VAS < 4.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to first dose of morphine administrated).
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded before skin incision, one minute after skin incision and then recorded regularly every 10 minutes.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded before skin incision, one minute after skin incision and then recorded regularly every 10 minutes.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 6, 8, 12, and 24 h postoperatively.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.